CLINICAL TRIAL: NCT07257198
Title: Evaluation of an asPirin-free Strategy With ticAgrelor in patieNTs witH a Myocardial Infarction treatEd Medically alONe (PANTHEON)
Brief Title: Aspirin-free Strategy With Ticagrelor in Patients With a Myocardial Infarction Treated Medically Alone
Acronym: PANTHEON
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Guillaume Marquis-Gravel, Associate professor of clinic, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-33-2026-3610; 202409PJT-525999-RC1-CFCK-1990 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: NSTEMI - Non-ST Segment Elevation MI; STEMI (ST Elevation MI); Myocardial Infarction
Keywords: Dual antiplatelet therapy; NSTEMI; medical treatment; STEMI; aspirin; ticagrelor; bleeding; ischemic events; randomized trial; pragmatic trial; randomized controlled trial
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Myocardial Infarction; Hemorrhage | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor monotherapy (Experimental): Ticagrelor 90 mg orally twice daily + placebo orally once daily
  Interventions: Drug: Ticagrelor + placebo
- DAPT with ticagrelor and aspirin (Active Comparator): Ticagrelor 90 mg orally twice daily + aspirin 80 mg orally once daily
  Interventions: Drug: Ticagrelor + aspirin

INTERVENTIONS:
Drug: Ticagrelor + placebo — Ticagrelor 90 mg twice daily + placebo once daily
  Arms: Ticagrelor monotherapy
Drug: Ticagrelor + aspirin — Ticagrelor 90 mg twice daily + aspirin 80 mg once daily
  Arms: DAPT with ticagrelor and aspirin

SUMMARY:
In patients with a myocardial infarction (MI) treated medically alone, the objective of the PANTHEON trial is to evaluate if ticagrelor monotherapy reduces bleeding events, without an increase in patient-oriented ischemic events, compared with standard dual antiplatelet therapy (DAPT) with aspirin and ticagrelor for 12 months.

DETAILED DESCRIPTION:
Coronary artery disease is associated with more than 9 million deaths per year worldwide. Following hospital discharge for an MI, both bleeding and recurrent ischemic events are associated with a high risk of subsequent mortality. However, the optimal antiplatelet strategy balancing bleeding and ischemic risks in the vulnerable population of patients with a medically managed MI patients (without revascularization) remains unknown, leading to substantial variability in clinical practice. This group represents 35-45% of patients wit hMI in Canada and the United States.

Primary Objectives To evaluate whether ticagrelor monotherapy is superior to dual antiplatelet therapy (DAPT) in reducing the risk of type 2, 3, or 5 bleeding events according to the BARC classification at 12 months.

To evaluate whether ticagrelor monotherapy is non-inferior to dual antiplatelet therapy (DAPT) for the composite endpoint of all-cause mortality, myocardial infarction, stroke, or coronary revascularization - a standardized, patient-centered ischemic clinical endpoint as defined by the Academic Research Consortium - at 12 months.

Secondary Objectives To evaluate differences between ticagrelor monotherapy and DAPT regarding the following endpoints at 12 months: individual components of the two primary endpoints; BARC type 3 or 5 bleeding; TIMI minor or major bleeding and its individual components; cardiovascular mortality; any coronary revascularization; the composite of all-cause mortality, MI, or stroke; and NACE, a composite of all-cause mortality, MI, stroke, any coronary revascularization, or type 2, 3, or 5 BARC bleeding.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years;
* Hospitalized for type 1 MI, according to the 4th Universal Definition of MI;
* Coronary angiogram performed;
* Planned for medical management alone, without revascularization;
* Willingness to participate and to attend study visits;
* Expected life expectancy ≥12 months.

Exclusion criteria:

* Patients hospitalized for type 2-5 MI, or unstable angina, according to the 4th Universal Definition of MI;
* Patients hospitalized for a STEMI with an acute thrombotic lesion of a major epicardial vessel;
* Elevations in cardiac biomarkers (troponins or CK-MB) that is believed by the investigator not to be of ischemic origin (e.g. myocardial injury, myocarditis, Takotsubo syndrome, etc.);
* Confirmed or suspected spontaneous coronary artery dissection;
* Concomitant indication for chronic oral anticoagulant;
* Concomitant non-coronary indication for dual antiplatelet therapy;
* Use of any non-trial antiplatelet drug that needs to be continued based on the judgement of the treating physician;
* Previous hospitalization for MI, PCI, or CABG within 12 months;
* Known hypersensitivity, intolerance, or contra-indication to ASA or ticagrelor;
* Unsuitability for either randomization treatment, based on the judgement of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2570 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding | From randomization to 12 months
  Time to first BARC type 2, 3, or 5 bleeding
Patient-oriented ischemic clinical endpoint | From randomization to 12 months
  Time to first composite of all-cause mortality, MI, stroke, or any coronary revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No